CLINICAL TRIAL: NCT01415453
Title: Evoked Visual Response Using Pulsed Ultrasound
Brief Title: Evoked Retinal Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Ronald H. Silverman, Professor of Ophthalmic Science, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AAAI1650
Record Dates: First submitted 2011-07-25; First posted 2011-08-12 (Estimated); Results first posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-03

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; acoustic radiation force ultrasound; RP; visual field loss; Photoreceptor; Vision loss; retina; progressive vision loss; ultrasound
MeSH Terms: conditions — Retinitis Pigmentosa; Vision Disorders | interventions — Ultrasonic Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retinitis Pigmentosa (Experimental): Subject will have retinitis pigmentosa and will be legally blind in one or both eyes
  Interventions: Procedure: Ultrasound Stimulus

INTERVENTIONS:
Procedure: Ultrasound Stimulus — Short pulses of focused ultrasound will be directed at spots on the retinal surface.
  Other Names: pulsed ultrasound

SUMMARY:
Retinitis pigmentosa (RP) is the name given to a group of inherited eye diseases that affect the retina (the light-sensitive part of the eye). RP causes the breakdown of photoreceptor cells (cells in the retina that detect light). Photoreceptor cells capture and process light helping us to see. As these cells breakdown and die, people experience progressive vision loss. There is no known cure for retinitis pigmentosa. The investigators have observed that short pulses of focused ultrasound can cause perception of light when directed to spots on the retinal surface. The investigators propose to conduct a study to determine if pulsed ultrasound will stimulate the perception of light in the absence of functional photoreceptors in people with RP

DETAILED DESCRIPTION:
Patients affected by retinitis pigmentosa (RP) and related diseases suffer loss of vision due to death of photoreceptor cells. The investigators have observed that short pulses of focused ultrasound can cause perception of light (phosphenes) when directed to spots on the retinal surface. If this phenomenon is caused by direct stimulation of the retinal nerves, which seems probable, then it might be possible to use this phenomenon to produce a form of vision in such patients. The investigators propose to conduct a study of a small cohort of patients affected by RP to determine if pulsed ultrasound will evoke a perception of light in the absence of functional photoreceptors.

ELIGIBILITY:
Inclusion Criteria:

* retinitis pigmentosa
* legally blind in at least one eye

Exclusion Criteria:

* unable to lay down on an exam table

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Silverman, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at the Department of Ophthalmology, Columbia University Medical Center from July 2011 to June 2012.
Pre-assignment Details: No significant events followed enrollment prior to group assignment. There was only one group in this study: people with retinitis pigmentosa who were legally blind.
Period: Overall Study
Arm/Group | Retinitis Pigmentosa
Started | 1
Imaging Study | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Retinitis Pigmentosa
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Phosphene Perception in Response to Ultrasound Pulse.
Description: The investigators will test the hypothesis that compression of retinal nerves by ultrasound force will cause perception of light (phosphenes) in blind subjects lacking functioning photoreceptors (retinitis pigmentosa). With each of two 5 msec ARFI exposures, if the subject either perceived the spark of light (phosphene), then it was documented as a positive response; if they did not, it was marked as a negative response.
Time Frame: Subjects will undergo a single examination of approximately 15 minute duration during which they will report perception of phosphenes during ultrasound exposure.
Population: Only one subject was examined.
Measure: Number; unit: participants
Arm/Group | Retinitis Pigmentosa
Number analyzed (Participants) | 1
participants
  Positive Evoked Response | 0
  Negative Evoked Response | 1

ADVERSE EVENTS:
Arm/Group | Retinitis Pigmentosa
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Difficulty in recruiting appropriate volunteers. Study terminated due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No